CLINICAL TRIAL: NCT04348591
Title: Identifying the Optimal Neural Target for Misophonia Interventions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Misophonia Research Fund (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: Pro00103863
Record Dates: First submitted 2020-04-07; First posted 2020-04-16 (Actual); Results first posted 2023-08-25 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Misophonia; Emotion Dysregulation
Keywords: neurostimulation; neuroscience; misophonia; emotion dysregulation; insula
MeSH Terms: conditions — misophonia | interventions — Cognitive Restructuring; Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: The investigators plan to compare adults who report misophonia with adults who report clinical emotional dysregulation in their neurobiological response to misophonic, aversive, and neutral sounds
Who Masked: Participant, Investigator
Masking Description: All participants will undergo different types of neurostimulation to probe different areas of the emotion regulation and misophonic networks while being exposed to sounds. One of these neurostimulation blocks will involve sham (inactive) neurostimulation. The investigator and the participants will be blind to which block has active and which block has sham neurostimulation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Misophonia Group (Experimental): Participants who endorse Misophonia will undergo a neuroimaging session to identify different neurostimulation targets. Then Misophonic participants will be exposed to aversive and neutral sounds while receiving real or sham neurostimulation over different pre-established neural targets.
  Interventions: Behavioral: Cognitive Restructuring; Device: neurostimulation
- Emotional Dysregulation Clinical Group (Active Comparator): Participants who self report high emotional dysregulation and who meet diagnostic criteria for a DSM disorder will undergo a neuroimaging session to identify different neurostimulation targets. Then these participants will be exposed to aversive and neutral sounds while receiving real or sham neurostimulation over different pre-established neural targets.
  Interventions: Behavioral: Cognitive Restructuring; Device: neurostimulation

INTERVENTIONS:
Behavioral: Cognitive Restructuring — All participants will learn how to change their thinking in order to be less upset when confronted with stressors
Device: neurostimulation — all participants will receive inhibitory, excitatory, and sham transcranial magnetic stimulation over different neural targets during the experimental session. The purpose of the neurostimulation is not treatment, but causal interference/enhancing of brain circuitry to identify candidate neural regions for future interventions
  Other Names: transcranial magnetic stimulation

SUMMARY:
Misophonia, the inability to tolerate certain repetitive aversive sounds that are common, is gaining recognition as a debilitating condition. It is not a well-understood condition and there are no known treatments. Up to one in five people report moderate or higher misophonia symptoms; nevertheless, resources aimed at understanding and treating this problem are scarce. In order to align misophonia research with the priorities of large funding agencies such as the National Institute of Mental Health, the investigators propose a novel study aimed at separating misophonic distress from other types of emotional distress. The investigators plan to examine changes in brain activation during presentation and regulation of misophonic versus distressing sounds. Emergent neural networks that may be involved in misophonia will then be tested in the lab with the use of noninvasive neurostimulation, a novel tool that can enhance or inhibit activation in a targeted brain region. The investigators plan to modulate activation in key areas of the misophonia brain circuitry with the aim to identify the optimal neural target for misophonia interventions. Our multidisciplinary team at the Duke Center for Misophonia and Emotion Regulation brings together experts in misophonia, neuroscience, neuromodulation, neurology, and biostatistics who share the long-term goal of developing and refining an intervention for this condition in an environment that is optimal to conduct the proposed research.

The investigators propose to recruit adults who self-report significant misophonia symptoms and adults who meet criteria for a current psychiatric disorder and who self-report difficulties calming down when upset. All participants will undergo a brain imaging session during which misophonic cues; distressing, non-misophonic cues; or neutral cues will be presented. Participants will then be asked to experience, or attempt to downregulate emotions associated with these cues. Based on the imaging results, two personalized neurostimulation targets will be identified: (1) the region in the frontal cortex with the most activity during the downregulation of misophonic versus neutral sounds and (2) the prefrontal region with the strongest functional connectivity to the anterior insular cortex. Participants will receive real or sham neurostimulation over the prefrontal cortex and insula in a random order, while engaging in listening to versus downregulating misophonic, aversive, or neutral cues. The investigators plan to assess emotional dysregulation, psychopathology, and misophonia with a multi-method battery of measures during all three study appointments. Feasibility and acceptability will be examined qualitatively. If successful, our study can be the first step in a series of investigations that establish the unique targets for neural intervention for misophonia.

DETAILED DESCRIPTION:
Consistent with NIMH strategic priorities, neural targets that account for individual differences are needed for the next generation of mental health interventions. Misophonia, the inability to tolerate certain aversive repetitive and common sounds, is gaining rapid recognition as a debilitating condition that is not currently well understood and for which interventions do not yet exist. In order to align research efforts to understand and treat misophonia with NIMH priorities, the investigators propose to conduct an experimental study that differentiates the neural circuitry of misophonia-induced distress from other types of emotional distress, and that begins to identify the optimal neural target for possible interventions. Noninvasive neurostimulation (i.e., the purposeful modulation of neural circuitry), such as repetitive transcranial magnetic stimulation (rTMS), is a powerful tool which can modulate neuronal activation and can be used to examine the responsiveness of neural circuits to intervention. Therefore, for this project, the investigators bring together a multidisciplinary team of researchers with expertise in misophonia, neuroscience, neuromodulation, biostatistics, and neurology with the aims to: (1) differentiate the brain circuitry dysfunction in misophonia compared to non-misophonia emotional distress and (2) identify the optimal intervention target for changing misophonic distress using rTMS. The investigators propose to recruit adults who self-report significant misophonia symptoms and a comparison group of adults who meet criteria for a current psychiatric disorder and who self-report high emotional dysregulation. Those who have contra-indications for MRI or rTMS will be excluded. All participants will undergo an MRI session during which misophonic cues; aversive, non-misophonic cues; or neutral cues will be presented. Participants will be asked to listen only or listen and attempt to downregulate emotions associated with these cues. Functional MRI (fMRI) analysis will then be performed to define two personalized neurostimulation targets defined as the region in the frontal cortex that is the most (1) activated during emotion regulation and (2) connected to the anterior insular cortex (AIC) during emotional experiencing. Participants will be assigned to receive active or sham neurostimulation over target 1 and target 2 in a random order, while engaged in listening to versus downregulating misophonic, aversive, or neutral cues. The investigators plan to employ excitatory neuromodulation to examine the effects of enhancing prefrontal cortex activation during emotion regulation. The investigators also plan to employ inhibitory neuromodulation to examine the effects of inhibiting AIC activation during listening only without efforts to regulate emotional distress. The investigators plan to assess emotional dysregulation, psychopathology, and misophonia with a multi-method battery of measures during all three study appointments. Feasibility and acceptability will be examined qualitatively. The investigators will use results from this study to design larger trials and to seek federal funding with the ultimate goal of designing an effective misophonia intervention. If successful, our study can be the first step in a series of investigations that establish the unique targets for neural intervention for misophonia.

ELIGIBILITY:
Interested participants will be excluded if:

1. current or past history of mania or psychosis,
2. verbal IQ < 70,
3. not medically cleared for TMS or fMRI (for example taking medications known to reduce the seizure threshold such as Lamictal, Lithium, Clozaril, stimulants including the ADHD medications (e.g. Ritalin, Adderall), Wellbutrin/Buproprion, Provigil (Modafinil), Aminophylline, and Theophylline, implants, TBI, stroke, etc),
4. going to jail in the next 2 months,
5. pregnant,
6. high risk for suicide
7. moderate/severe current alcohol or substance dependence,
8. cannot come to Duke for the three study visits.

Inclusion criteria are:

1. stable psychotherapy and medication for at least 4 weeks
2. self reports high emotional dysregulation OR misophonia

Participants will be matched on gender and age between the two groups

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2020-10-28 (Actual); Primary Completion 2022-05-27 (Actual); Study Completion 2022-05-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrada D Neacsiu, PhD, Principal Investigator — Duke Health
Locations (1):
- Duke University Medical Center-Civitan Bldg, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Participant data from the study was shared to the Duke Research Data Repository (RDR).
  Neacsiu, A., LaBar, K., Rosenthal, M. Z., Bukhari-Parlakturk, N., Kelley, L. (2022). Identifying the optimal neural target for misophonia interventions. Duke Research Data Repository. https://doi.org/10.7924/r4ww7jg4k
Time Frame: Data in SPSS and .csv format along with the data dictionary was submitted and accepted on 10/27/2022. It is available currently at the Duke Research Data Repository (RDR). The Duke RDR provides access to and preservation of the data for a minimum period of 25 years.
Access Criteria: Open to any researcher to view and access.
URL: https://doi.org/10.7924/r4ww7jg4k

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through online websites (e.g., Craigslist, Dukelist), social media (Facebook, Instagram, Reddit), flyers, and electronic medical record outreach. Participants reached the study predominantly by seeing advertisements on social media and research websites. Many participants who met the severity cutoff for misophonia also found the study via self-guided internet search.
Pre-assignment Details: Top reasons for not qualifying included emotion dysregulation & misophonia severity too low; too low severity for misophonic group, but too many misophonic symptoms for control group; moderate/severe current alcohol or substance use disorder; TMS/MRI contraindications; or could not provide usable MRI data.
Groups:
- Misophonia Group: Participants who endorse Misophonia will undergo a neuroimaging session to identify different neurostimulation targets. Then Misophonic participants will be exposed to misophonic, aversive and neutral sounds while receiving real or sham neurostimulation over different pre-established neural targets.
  Cognitive Restructuring: All participants will learn how to change their thinking in order to be less upset when confronted with stressors
  neurostimulation: all participants will receive inhibitory, excitatory, and sham transcranial magnetic stimulation over different neural targets during the experimental session. The purpose of the neurostimulation is not treatment, but causal interference/enhancing of brain circuitry to identify candidate neural regions for future interventions
- Emotional Dysregulation Clinical Group: Participants who self report high emotional dysregulation and who meet diagnostic criteria for a DSM disorder will undergo a neuroimaging session to identify different neurostimulation targets. Then these participants will be exposed to misophonic, aversive and neutral sounds while receiving real or sham neurostimulation over different pre-established neural targets.
  Cognitive Restructuring: All participants will learn how to change their thinking in order to be less upset when confronted with stressors
  neurostimulation: all participants will receive inhibitory, excitatory, and sham transcranial magnetic stimulation over different neural targets during the experimental session. The purpose of the neurostimulation is not treatment, but causal interference/enhancing of brain circuitry to identify candidate neural regions for future interventions
Period: Imaging Session (120 Min)
Arm/Group | Misophonia Group | Emotional Dysregulation Clinical Group
Started | 29 | 30
Completed | 27 | 27
Not Completed | 2 | 3
Not completed — Lost to Follow-up | 0 | 2
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 2 | 0
Period: CR Training (45 Min)
Arm/Group | Misophonia Group | Emotional Dysregulation Clinical Group
Started | 27 | 27
Completed | 27 | 27
Not Completed | 0 | 0
Period: Experimental Task (45 Min)
Arm/Group | Misophonia Group | Emotional Dysregulation Clinical Group
Started | 27 | 27
Completed Sham rTMS Experimental Condition (Each participant listened to neutral, aversive, and misophonic trigger sounds that were personalized while receiving sham neurostimulation) | 26 | 27
Completed HF rTMS Over the Right dlPFC Experimental Condition (Each participant listened to neutral, aversive, and misophonic trigger sounds that were personalized while receiving high frequency neurostimulation over the right dlPFC) | 26 | 27
Completed LF rTMS Over the Right mPFC Experimental Condition (Each participant listened to neutral, aversive, and misophonic trigger sounds that were personalized while receiving low frequency neurostimulation over the right mPFC) | 27 | 27
Completed | 27 | 27
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Misophonia Group | Emotional Dysregulation Clinical Group | Total
Number analyzed (Participants) | 29 | 30 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.59 (9.79) | 27.07 (8.28) | 28.31 (9.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 26 | 52
  Male | 3 | 4 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 7 | 8
  Not Hispanic or Latino | 28 | 23 | 51
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 10 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 28 | 17 | 45
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 29 | 30 | 59
misophonia questionnaire Subscale 1 [Mean (Standard Deviation); unit: units on a scale] — Trigger Subscale 1 of the misophonia questionnaire includes 8 triggers that participants rate they are sensitive to on a scale of 0 to 4 where 0=Not at all true to 4=Always True. A total subscale score is computed by averaging the items (range 0-4). Higher score indicates higher misophonia sensitivity (i.e., more severity).
  units on a scale | 2.86 (0.43) | 1.37 (0.87) | 2.10 (1.02)
misophonia questionnaire Subscale 2 [Mean (Standard Deviation); unit: units on a scale] — Response Subscale 2 of the Misophonia questionnaire has 11 potential statements that participants rate occur when triggered on a scale of 0 to 4 where 0=Never to 4=Always. A total subscale score is computed by averaging the scores on these items. Higher scores indicate more misophonia severity.
  units on a scale | 2.83 (0.38) | 1.08 (0.69) | 1.97 (1.04)
misophonia questionnaire severity [Mean (Standard Deviation); unit: units on a scale] — 1 question where participants rate the severity of their sound sensitivity from 1=minimal to 15=very severe.
  units on a scale | 9.18 (1.63) | 3.45 (2.47) | 6.26 (3.56)
Difficulties in emotion regulation scale [Mean (Standard Deviation); unit: units on a scale] — Difficulties with emotion regulation statements were rated on frequency on a scale of 1 to 5 where 1=Almost Never and 5=Almost Always. After collecting the ratings, in scoring some of the items on the scale are reverse scored. Next, a score is computed by adding all the items on the scale, yielding a total score that ranges from 36 to 180. Higher scores indicate more difficulties with emotional dysregulation.
  units on a scale | 108.16 (24.69) | 117.17 (16.39) | 112.83 (21.11)

OUTCOME MEASURES:

1. Primary Outcome: Physiological Outcome: High Frequency Heart Rate Variability (HF-HRV) Recorded During Experimental Blocks
Description: HF-HRV was extracted from 2 minute blocks during which participants engage in a behavioral strategy (listen or downregulate emotions using cognitive restructuring), while listening to neutral, aversive, and misophonic sounds and receive active or sham neurostimulation. The results represent the average HF-HRV during experimental blocks. The raw values were transformed using a logarithmic function to preserve the normality assumption.
Time Frame: Two minute blocks during the neurostimulation experimental session during which participants listened to or downregulated emotions associated with experimental sounds (45 minutes total).
Population: Participants who completed the study.
Measure: Mean (Standard Deviation); unit: lg(ms^2)
Arm/Group | Misophonia Group | Emotional Dysregulation Clinical Group
Number analyzed (Participants) | 27 | 27
lg(ms^2)
  listen to neutral sound+ sham stimulation: number analyzed (Participants) | 26 | 27
  listen to neutral sound+ sham stimulation | 1.8903 (.49961) | 1.9422 (.51434)
  listen to a neutral sound+ HF rTMS stimulation: number analyzed (Participants) | 26 | 27
  listen to a neutral sound+ HF rTMS stimulation | 1.9420 (.47814) | 1.9465 (.52974)
  listen to a neutral sound+ LF rTMS | 1.8923 (.4136) | 1.9771 (.61184)
  listen to an aversive sound+sham stimulation: number analyzed (Participants) | 26 | 27
  listen to an aversive sound+sham stimulation | 1.9172 (.44301) | 1.9151 (.49276)
  listen to an aversive sound+ HF rTMS: number analyzed (Participants) | 26 | 27
  listen to an aversive sound+ HF rTMS | 1.9753 (.45907) | 2.0791 (.58066)
  listen to an aversive sound + LF rTMS | 1.8942 (.44218) | 1.9590 (.62018)
  listen to a misophonic sound + sham stimulation: number analyzed (Participants) | 26 | 27
  listen to a misophonic sound + sham stimulation | 1.8920 (.44746) | 1.8868 (.58837)
  listen to a misophonic sound + HF rTMS: number analyzed (Participants) | 26 | 27
  listen to a misophonic sound + HF rTMS | 1.9680 (.43347) | 2.0457 (.55137)
  listen to a misophonic sound + LF rTMS | 1.8289 (.48734) | 1.9392 (.61046)
  downregulate emotions during aversive sounds + sham stimulation: number analyzed (Participants) | 26 | 27
  downregulate emotions during aversive sounds + sham stimulation | 1.9216 (.46655) | 1.9390 (.61942)
  downregulate emotions during aversive sounds + HF rTMS: number analyzed (Participants) | 26 | 27
  downregulate emotions during aversive sounds + HF rTMS | 1.9319 (.45462) | 2.0262 (.55149)
  downregulate emotions during aversive sounds + LF rTMS | 1.8740 (.45462) | 1.9669 (.64162)
  downregulate emotions during misophonic sounds + sham stimulation: number analyzed (Participants) | 26 | 27
  downregulate emotions during misophonic sounds + sham stimulation | 1.9290 (.47660) | 1.9362 (.56408)
  downregulate emotions during misophonic sounds + HF rTMS: number analyzed (Participants) | 26 | 27
  downregulate emotions during misophonic sounds + HF rTMS | 1.9259 (.46639) | 1.9962 (.57097)
  downregulate emotions during misophonic sounds + LF rTMS | 1.8882 (.48890) | 1.9281 (.58576)
Statistical Analysis 1: Comparison: Misophonia Group vs Emotional Dysregulation Clinical Group; A MMANOVA analysis using an unstructured covariance structure examined main effects of experimental group, instruction provided, headache, racial background, and type of neurostimulation administered. HF-HRV was transformed using an lg function for normality; Test type: Superiority; p = .221, Mixed Models Analysis — This p value corresponds to the main effect for experimental group; a-priori threshold was .012; Mean Difference (Final Values) = -.046, 95% CI 2-sided [-.12 to .029], Standard Error of Mean .037
Statistical Analysis 2: Comparison: Misophonia Group vs Emotional Dysregulation Clinical Group; A MMANOVA analysis using an unstructured covariance examined the main effect of type of neurostimulation provided; Test type: Superiority — This is a within subject analysis that uses data across groups, controlling for the effect of neurostimulation alone, coil to cortex distance, and racial background; p = .008, Mixed Models Analysis; Comparison between sham neurostimulation and high frequency neurostimulation; Mean Difference (Final Values) = .059, 95% CI 2-sided [.016 to .103], Standard Error of Mean .022
Statistical Analysis 3: Comparison: Misophonia Group vs Emotional Dysregulation Clinical Group; A MMANOVA analysis using an unstructured covariance structure examined the main effect of type of neurostimulation provided; Test type: Superiority — The analysis controls for coil to cortex distance, racial background and effect of neurostimulation alone. It compares sham stimulation with low frequency neurostimulation; p = .001, Mixed Models Analysis; Mean Difference (Final Values) = .07, 95% CI 2-sided [.029 to .111], Standard Error of Mean .021

2. Primary Outcome: Skin Conductance Level (SCL)
Description: Physiological arousal measured by SCL during each experimental block was extracted using Acqknowledge software and BIOPAC hardware (during the neurostimulation session). Raw galvanic skin response was continuously collected throughout the experiment. Raw data was then examined for abrupt changes (skin conductance responses), which were removed. The processed data was then averaged for each two minute experimental block. Higher SCL means higher arousal.
Time Frame: Two minute blocks during the neurostimulation experimental session (when participants listened to or downregulated emotions associated with experimental sounds)
Population: Participants who completed the study.
Measure: Mean (Standard Deviation); unit: microsemens
Arm/Group | Misophonia Group | Emotional Dysregulation Clinical Group
Number analyzed (Participants) | 27 | 27
microsemens
  listen to neutral sounds + sham stimulation: number analyzed (Participants) | 26 | 27
  listen to neutral sounds + sham stimulation | 8.42392 (3.228892) | 8.90082 (5.259539)
  listen to neutral sounds + HF rTMS: number analyzed (Participants) | 26 | 27
  listen to neutral sounds + HF rTMS | 8.51538 (3.820940) | 9.30579 (5.232129)
  listen to neutral sounds + LF rTMS | 8.39378 (3.569227) | 8.83644 (5.731341)
  listen to aversive sounds + sham stimulation: number analyzed (Participants) | 26 | 27
  listen to aversive sounds + sham stimulation | 9.18323 (3.275174) | 9.40404 (5.249783)
  listen to aversive sounds + HF rTMS: number analyzed (Participants) | 26 | 27
  listen to aversive sounds + HF rTMS | 9.56538 (4.100446) | 10.45648 (5.395880)
  listen to aversive sounds + LF rTMS | 9.41889 (3.675953) | 9.51379 (5.677760)
  listen to misophonic sounds + sham stimulation: number analyzed (Participants) | 26 | 27
  listen to misophonic sounds + sham stimulation | 8.83446 (3.160085) | 9.17171 (5.249371)
  listen to misophonic sounds + HF rTMS: number analyzed (Participants) | 26 | 27
  listen to misophonic sounds + HF rTMS | 8.68612 (3.446615) | 9.68599 (5.220985)
  listen to misophonic sounds + LF rTMS | 8.89759 (3.950378) | 8.85123 (5.617469)
  downregulate distress associated with aversive sounds+ sham stimulation: number analyzed (Participants) | 26 | 27
  downregulate distress associated with aversive sounds+ sham stimulation | 8.5036 (3.5264) | 8.88481 (5.501042)
  downregulate distress associated with aversive sounds+ HF rTMS: number analyzed (Participants) | 26 | 27
  downregulate distress associated with aversive sounds+ HF rTMS | 8.51065 (3.714333) | 9.53835 (5.269438)
  downregulate distress associated with aversive sounds+ LF rTMS | 8.34333 (3.567143) | 8.82512 (5.850350)
  downregulate distress associated with misophonic sounds+ sham stimulation: number analyzed (Participants) | 26 | 27
  downregulate distress associated with misophonic sounds+ sham stimulation | 8.66058 (3.438065) | 8.64721 (5.321361)
  downregulate distress associated with misophonic sounds+ HF rTMS: number analyzed (Participants) | 26 | 27
  downregulate distress associated with misophonic sounds+ HF rTMS | 8.38327 (3.611908) | 9.37240 (5.049701)
  downregulate distress associated with misophonic sounds+ LF rtMS | 8.43874 (3.658122) | 8.82144 (5.888309)
Statistical Analysis 1: Comparison: Misophonia Group vs Emotional Dysregulation Clinical Group; A MMANOVA analysis using an unstructured covariance structure examined changes in SCL between groups, experimental types of neurostimulation, and their interaction, controlling for baseline, racial background, coil to cortex distance, and headache; Test type: Superiority; p = .34, Mixed Models Analysis; Mean Difference (Final Values) = .223, 95% CI 2-sided [-.243 to .689], Standard Error of Mean .232 — This is the result for the main effect found of group (emotion dysregulation group versus misophonia)
Statistical Analysis 2: Comparison: Misophonia Group vs Emotional Dysregulation Clinical Group; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = .001, Mixed Models Analysis; This is the main effect of neurostimulation condition. Specifically here we show the difference in estimated marginal means between sham and HF-rTMS; Mean Difference (Final Values) = .493, 95% CI 2-sided [.198 to .787], Standard Error of Mean .148
Statistical Analysis 3: Comparison: Misophonia Group vs Emotional Dysregulation Clinical Group; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = .002, Mixed Models Analysis; This is the main effect of neurostimulation administered, specifically comparing estimated marginal means for sham and LF-rTMS; Mean Difference (Final Values) = .469, 95% CI 2-sided [.182 to .757], Standard Error of Mean .144
Statistical Analysis 4: Comparison: Misophonia Group vs Emotional Dysregulation Clinical Group; The investigators tested the interaction between experimental neurostimulation (sham, active high frequency rTMS, active low frequency rTMS), instruction provided (listen to neutral sound; listen to aversive sound, listen to misophonic sound, downregulate aversive sound, downregulate misophonic sound), and group (misophonic, clinical control) as part of the same MMANOVA analysis described above (i.e., controlling for coil-to-cortex distance, racial background, baseline, & presence of headache); Test type: Superiority; p = .0005, Mixed Models Analysis; Mean Difference (Final Values) = 0.73 — mean difference between sham and HF-rTMS for misophonia participants only when downregulating misophonic sounds

3. Primary Outcome: Behavioral Outcome: Acceptability of Procedures
Description: The investigators will record how many participants completed the neurostimulation session as a marker of acceptability.
Time Frame: At the end of the neurostimulation session (session 3 in the experiment), which occured within a month of the initial assessment
Population: Participants who completed the study
Measure: Count of Participants; unit: Participants
Arm/Group | Misophonia Group | Emotional Dysregulation Clinical Group
Number analyzed (Participants) | 27 | 27
Participants | 27 | 27

4. Primary Outcome: Neuroimaging Outcome: Differential Change in BOLD Signal Between Groups Within the Dorsolateral Prefrontal Cortex (dlPFC), That is Greater During Regulation of Misophonic Versus Non-misophonic Distress
Description: Blood Oxygenation Level Dependent (BOLD) imaging is a technique that is commonly used for estimating brain activity using functional magnetic resonance imaging (fMRI). Change in the fMRI BOLD signal notes changes in brain blood flow and blood oxygenation, which are associated with neuronal activity. Higher values indicate higher activity changes within a contrast of interes. A dlPFC mask was employed to find the maximum value of the [downregulate misophonic sounds > downregulate aversive sounds] contrast in this region. Once the voxel containing this maximum was identified, a 6 mm sphere ROI was created around this spot (restricted to the dlPFC mask) and the average contrast value within this sphere was used as the outcome variable.
Time Frame: during the neuroimaging session, within a month of the intake assessment
Population: Participants who completed the study.
Measure: Mean (Standard Deviation); unit: BOLD arbitrary units
Arm/Group | Misophonia Group | Emotional Dysregulation Clinical Group
Number analyzed (Participants) | 27 | 27
BOLD arbitrary units | .4572 (.58605) | .4288 (.32026)
Statistical Analysis 1: Comparison: Misophonia Group vs Emotional Dysregulation Clinical Group; An independent samples t-test was conducted to examine differences between groups in BOLD bilateral dlPFC signal during the regulation of misophonic versus aversive sounds. One outlier was removed from the misophonia group to avoid violating the normality assumption; Test type: Superiority; p = .57, t-test, 2 sided; Mean Difference (Final Values) = .0563, 95% CI 2-sided [-.14149 to .25411], Standard Error of Mean .09853

5. Primary Outcome: Neuroimaging Outcome: Differential Change in BOLD Signal Within the Ventromedial Prefrontal Cortex (vmPFC) When Engaging in the Regulation of Emotional Versus Misophonic Distress
Description: Blood Oxygenation Level Dependent (BOLD) imaging is a technique that is commonly used for estimating brain activity using functional magnetic resonance imaging (fMRI). Change in the fMRI BOLD signal notes changes in brain blood flow and blood oxygenation, which are associated with neuronal activity. A vmPFC mask was employed to find the maximum value of the [downregulate misophonic sounds > downregulate aversive sounds] contrast in this region. Once the voxel containing this maximum was identified, a 6 mm sphere ROI was created around this spot (restricted to the vmPFC mask) and the average contrast value within this sphere will be used as the outcome variable. Higher scores indicate more activity when downregulating misophonic versus aversive sounds.
Time Frame: during the neuroimaging session, within a month of the intake assessment
Population: Participants who completed the study.
Measure: Mean (Standard Deviation); unit: BOLD arbitrary units
Arm/Group | Misophonia Group | Emotional Dysregulation Clinical Group
Number analyzed (Participants) | 27 | 27
BOLD arbitrary units | .4967 (.61469) | .5233 (.60430)
Statistical Analysis 1: Comparison: Misophonia Group vs Emotional Dysregulation Clinical Group; An independent samples t-test was conducted to examine differences between groups in vmPFC activation that was greater when downregulating misophonic versus non-misophonic distress. One participant from each group was excluded for being an outlier; Test type: Superiority; p = .778, t-test, 2 sided; 50 degrees of freedom; Mean Difference (Final Values) = 0.037293, 95% CI 2-sided [-0.226670 to 0.301257], Standard Error of Mean 0.131419

6. Primary Outcome: Neuroimaging Outcome: Differential Change in BOLD Signal Within the Anterior Insular Cortex (AIC) Activation When Being Presented With Cues for Emotional Versus Misophonic Distress
Description: Blood Oxygenation Level Dependent (BOLD) imaging is a technique that is commonly used for estimating brain activity using functional magnetic resonance imaging (fMRI). Change in the fMRI BOLD signal notes changes in brain blood flow and blood oxygenation, which are associated with neuronal activity. An AIC mask was employed to find the maximum value of the [hear misophonic sounds > hear aversive sounds] contrast in this region. Once the voxel containing this maximum was identified, a 6 mm sphere ROI was created around this spot (restricted to the AIC mask) and the average contrast value within this sphere will be used as the outcome variable. A larger score indicates more activity when hearing misophonic versus aversive sounds.
Time Frame: during the neuroimaging session, within a month of the intake assessment
Population: Participants who completed the study.
Measure: Mean (Standard Deviation); unit: BOLD arbitrary units
Arm/Group | Misophonia Group | Emotional Dysregulation Clinical Group
Number analyzed (Participants) | 27 | 27
BOLD arbitrary units | .3744 (.22996) | .3093 (.22876)
Statistical Analysis 1: Comparison: Misophonia Group vs Emotional Dysregulation Clinical Group; Mixed effects (FSL's FLAME 1; Oxford Univ., UK) whole brain analyses using cluster correction following a voxel-wise Z-score threshold of 2.3; Test type: Superiority; p < .05, mixed effects whole-brain using cluster; z score = 4.69

7. Secondary Outcome: Change in Subjective Units of Distress (SUDS)
Description: Self reported distress after experimental blocks will also be examined for differences when accounting for baseline distress (during the neurostimulation session). SUDS will be measured using a 0-9 sale, where 0 indicates no distress, and 9 indicates extreme distress. The outcome measure represents SUDS after negative sound presentations (misophonic and aversive) minus SUDS after baseline. Higher SUDS represents higher distress.
Time Frame: Baseline, during the experimental blocks during the neurostimulation session (which will occur within a month of the initial assessment)
Population: Participants who completed the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Misophonia Group | Emotional Dysregulation Clinical Group
Number analyzed (Participants) | 27 | 27
units on a scale
  listen to neutral sounds + sham stimulation: number analyzed (Participants) | 26 | 27
  listen to neutral sounds + sham stimulation | 0.2981 (1.35732) | 0.5370 (1.25621)
  listen to neutral sounds + HF rTMS: number analyzed (Participants) | 26 | 27
  listen to neutral sounds + HF rTMS | -0.5769 (1.45277) | -0.3611 (1.97866)
  listen to neutral sounds + LF rTMS | -0.2130 (1.61795) | 0.3056 (1.33576)
  listen to aversive sounds + sham stimulation: number analyzed (Participants) | 26 | 27
  listen to aversive sounds + sham stimulation | 1.3107 (1.94548) | 2.8795 (2.18199)
  listen to aversive sounds + HF rTMS: number analyzed (Participants) | 26 | 27
  listen to aversive sounds + HF rTMS | 0.6019 (2.11131) | 1.8505 (2.21404)
  listen to aversive sounds + LF rTMS | 0.8981 (1.66851) | 2.5463 (2.25224)
  listen to misophonic sounds + sham stimulation: number analyzed (Participants) | 26 | 27
  listen to misophonic sounds + sham stimulation | 4.4712 (2.38505) | 2.3426 (2.02398)
  listen to misophonic sounds+ HF rTMS: number analyzed (Participants) | 26 | 27
  listen to misophonic sounds+ HF rTMS | 3.3269 (2.71079) | 0.9815 (2.28764)
  listen to misophonic sounds + LF rTMS | 3.7037 (2.64490) | 1.9252 (1.98438)
  downregulate distress associated with aversive sounds+ sham stimulation: number analyzed (Participants) | 26 | 27
  downregulate distress associated with aversive sounds+ sham stimulation | 0.7184 (1.59913) | 1.3148 (1.29448)
  downregulate distress associated with aversive sounds+ HF rTMS: number analyzed (Participants) | 26 | 27
  downregulate distress associated with aversive sounds+ HF rTMS | -0.0288 (1.56079) | 0.1574 (1.74636)
  downregulate distress associated with aversive sounds+ LF rTMS | 0.2685 (1.27965) | 1.0926 (1.38441)
  downregulate distress associated with misophonic sounds+ sham stimulation: number analyzed (Participants) | 26 | 27
  downregulate distress associated with misophonic sounds+ sham stimulation | 3.3173 (2.45845) | 1.0472 (1.35494)
  downregulate distress associated with misophonic sounds+ HF rTMS: number analyzed (Participants) | 26 | 27
  downregulate distress associated with misophonic sounds+ HF rTMS | 2.0673 (2.70298) | -0.2963 (1.49303)
  downregulate distress associated with misophonic sounds+ LF rTMS | 2.50000 (2.71548) | 0.7778 (1.38977)
Statistical Analysis 1: Comparison: Misophonia Group vs Emotional Dysregulation Clinical Group; The MMANOVA analysis of SUDS used a Toeplitz covariance structure. The outcome variable was the difference between SUDS after each sound presentation and baseline, controlling for racial background, headache, and coil to cortex difference. Two participants were excluded from this analysis, one in each condition, because they provided outlier data; Test type: Superiority; p = .49, Mixed Models Analysis; This is the main effect from the MMANOVA analysis for group difference; Mean Difference (Final Values) = -.197, 95% CI 2-sided [-.766 to .372], Standard Error of Mean .283
Statistical Analysis 2: Comparison: Misophonia Group vs Emotional Dysregulation Clinical Group; The MMANOVA analysis of SUDS used a Toeplitz covariance structure. This analysis presents the main effect of neurostimulation experimental condition. The outcome variable was the difference between SUDS after each sound presentation and baseline, controlling for racial background, headache, and coil to cortex difference. Two participants were excluded from this analysis, one in each condition, because they provided outlier data; Test type: Superiority; p < .0000001, Mixed Models Analysis — This p-value corresponds to the difference between sham and HF-rTMS stimulation; Mean Difference (Final Values) = .909, 95% CI 2-sided [.62 to 1.97], Standard Error of Mean .147
Statistical Analysis 3: Comparison: Misophonia Group vs Emotional Dysregulation Clinical Group; [analysis description as in outcome 7, analysis 2]; Test type: Superiority; p = .018, Mixed Models Analysis — The test corresponds to the difference between sham and LF-rTMS; Mean Difference (Final Values) = .331, 95% CI 2-sided [.057 to .605], Standard Error of Mean .139
Statistical Analysis 4: Comparison: Misophonia Group vs Emotional Dysregulation Clinical Group; The MMANOVA analysis of SUDS used a Toeplitz covariance structure. This analysis presents the interaction effect of group by neurostimulation experimental condition. The outcome variable was the difference between SUDS after each sound presentation and baseline, controlling for racial background, headache, and coil to cortex difference. Two participants were excluded from this analysis, one in each condition, because they provided outlier data; Test type: Superiority; p < .000001, Mixed Models Analysis; Mean Difference (Final Values) = 1.02 — For participants with misophonia difference in distress produced by a misophonic sound when downregulating misophonic sounds while receiving sham vs.HF-rTMS

8. Secondary Outcome: Emotional Dysregulation as Measured by the Difficulties in Emotion Regulation Scale (DERS)
Description: A self report assessing difficulties regulating emotions will be examined before and after the experiment (i.e., at the end of the neurostimulation session). The DERS ranges from 36 to 180, with higher scores indicating more dysregulation.
Time Frame: From baseline to the end of neurostimulation session, an average of 4 weeks.
Population: Some participants dropped out or were lost to contact by follow up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Misophonia Group | Emotional Dysregulation Clinical Group
Number analyzed (Participants) | 29 | 30
score on a scale
  Baseline | 93.04 (21.17) | 112.43 (16.42)
  End of neurostimulation session: number analyzed (Participants) | 27 | 26
  End of neurostimulation session | 88.70 (21.76) | 99.85 (17.75)
Statistical Analysis 1: Comparison: Misophonia Group vs Emotional Dysregulation Clinical Group; Repeated measures ANOVA (controlling for racial background); Test type: Superiority; p < .001, ANCOVA — This is the result corresponding to the main effect of time in the repeated measures ANCOVA; Mean Difference (Final Values) = 9.53, Standard Error of Mean 1.92
Statistical Analysis 2: Comparison: Misophonia Group vs Emotional Dysregulation Clinical Group; Repeated measures ANOVA (controlling for racial background); Test type: Superiority; p > .012, ANCOVA; This analysis corresponds to the main effect of group

9. Secondary Outcome: Self-reported Health Status as Measured by the Patient Reported Outcome Measurement Information System (PROMIS)-43 Adult Profile
Description: The PROMIS-43 is a 43-item questionnaire assessing health status in seven domains: physical function, anxiety, depression, fatigue, sleep disturbance, pain interference, and participation in social roles. Lower scores indicate less impairment in functioning when compared to higher scores. Each item has five response options ranging in value from 1 to 5, except for the 1 Pain Intensity item which has eleven response options ranging in value from 0 to 10. A raw score is created from each domain that makes up the Profile. Each domain raw score ranging from 6-30 corresponds to a T-Score in the PROMIS scoring manual.
Time Frame: At baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Misophonia Group | Emotional Dysregulation Clinical Group
Number analyzed (Participants) | 29 | 30
score on a scale
  P43 Anxiety | 14.10 (5.37) | 13.70 (5.73)
  P43 Depression | 11.28 (6.05) | 13.03 (6.49)
  P43-Fatigue | 14.97 (7.27) | 15.80 (6.27)
  P43- Sleep disturbance | 13.24 (6.26) | 15.30 (4.83)
  P43- Ability to partake in social roles | 23.86 (4.60) | 23.07 (5.66)
  P43-Pain interference | 7.59 (3.09) | 7.93 (3.11)
  P43-Physical functioning | 29.76 (3.11) | 28.73 (2.36)
Statistical Analysis 1: Comparison: Misophonia Group vs Emotional Dysregulation Clinical Group; An independent samples t-test was conducted to examine between group differences at the intake assessment on the PROMIS Anxiety subscale; Test type: Superiority; p = .78, t-test, 2 sided
Statistical Analysis 2: Comparison: Misophonia Group vs Emotional Dysregulation Clinical Group; An independent samples t-test was conducted to examine between group differences at the intake assessment on the PROMIS Depression subscale; Test type: Superiority; p = .29, t-test, 2 sided
Statistical Analysis 3: Comparison: Misophonia Group vs Emotional Dysregulation Clinical Group; An independent samples t-test was conducted to examine between group differences at the intake assessment on the PROMIS Fatigue subscale; Test type: Superiority; p = .64, t-test, 2 sided
Statistical Analysis 4: Comparison: Misophonia Group vs Emotional Dysregulation Clinical Group; An independent samples t-test was conducted to examine between group differences at the intake assessment on the PROMIS Sleep disturbance subscale; Test type: Superiority; p = .16, t-test, 2 sided
Statistical Analysis 5: Comparison: Misophonia Group vs Emotional Dysregulation Clinical Group; An independent samples t-test was conducted to examine between group differences at the intake assessment on the PROMIS Ability to partake in social roles subscale; Test type: Superiority; p = .56, t-test, 2 sided

10. Secondary Outcome: Number of Clusters Across the Whole Brain With Significant BOLD Changes Between Groups When Contrasting the Exposure to Aversive Versus Neutral Sounds.
Description: Blood Oxygenation Level Dependent (BOLD) imaging is a technique that is commonly used for estimating brain activity using functional magnetic resonance imaging (fMRI). Change in the fMRI BOLD signal notes changes in brain blood flow and blood oxygenation, which are associated with neuronal activity. The BOLD signal contrast between engaging with aversive sounds and engaging with neutral sounds were compared between groups across the whole brain on a voxel-wise basis. Voxel-wise significant results (i.e., z > 2.3) were clustered to statistically correct for multiple comparisons. The number of significant clusters that emerged from this analysis in each group are presented as outcome.
Time Frame: During the neuroimaging session, within a month of the intake assessment
Measure: Number; unit: clusters where differences emerged
Arm/Group | Misophonia Group | Emotional Dysregulation Clinical Group
Number analyzed (Participants) | 29 | 30
clusters where differences emerged | 0 | 0

11. Secondary Outcome: Number of Clusters Across the Whole Brain With Significant BOLD Changes Between Groups When Contrasting the Exposure to Misophonic Versus Aversive Sounds.
Description: Blood Oxygenation Level Dependent (BOLD) imaging is a technique that is commonly used for measuring brain activity using functional magnetic resonance imaging (fMRI). Change in a BOLD signal detected in fMRI, notes changes in brain blood flow and blood oxygenation. Neural activation across the brain when engaging with misophonic sounds versus aversive sounds during the neuroimaging day. The BOLD signal contrast between engaging with misophonic sounds and engaging with aversive sounds were compared between groups across the whole brain on a voxel-wise basis. Voxel-wise significant results (i.e., z > 2.3) were clustered to statistically correct for multiple comparisons. The number of significant clusters that emerged from this analysis in each group are presented as outcome.
Time Frame: during the neuroimaging session, within a month of the intake assessment
Measure: Number; unit: clusters
Arm/Group | Misophonia Group | Emotional Dysregulation Clinical Group
Number analyzed (Participants) | 29 | 30
clusters | 6 | 3

12. Secondary Outcome: Number of Clusters Across the Whole Brain With Significant BOLD Changes Between Groups When Contrasting the Downregulation of Distress Associated With Misophonic Sounds to Exposure to Misophonic Sounds
Description: Blood Oxygenation Level Dependent (BOLD) imaging is a technique that is commonly used for estimating brain activity using functional magnetic resonance imaging (fMRI). Change in the fMRI BOLD signal notes changes in brain blood flow and blood oxygenation, which are associated with neuronal activity. The BOLD signal contrast between regulating versus engaging with misophonic sounds across the entire brain was compared between participant groups on a voxel-wise basis. Voxel-wise results were clustered to statistically correct for multiple comparisons. The number of significant clusters within each group are presented as outcome (more cluster indicates more differences during regulation in that group versus the control group).
Time Frame: during the neuroimaging session, within a month of the intake assessment
Measure: Number; unit: clusters
Arm/Group | Misophonia Group | Emotional Dysregulation Clinical Group
Number analyzed (Participants) | 29 | 30
clusters | 1 | 0

13. Secondary Outcome: Number of Clusters Across the Whole Brain With Significant BOLD Changes Between Groups When Contrasting the Downregulation of Distress Associated With Aversive Sounds to Exposure to AversiveSounds
Description: Blood Oxygenation Level Dependent (BOLD) imaging is a technique that is commonly used for estimating brain activity using functional magnetic resonance imaging (fMRI). Change in the fMRI BOLD signal notes changes in brain blood flow and blood oxygenation, which are associated with neuronal activity. The BOLD signal contrast between regulating and engaging with aversive sounds was compared between participant groups on a voxel-wise basis. Voxel-wise results were clustered to statistically correct for multiple comparisons. The number of significant clusters within each group are reported as the outcome measure.
Time Frame: during the neuroimaging session, within a month of the intake assessment
Measure: Number; unit: clusters
Arm/Group | Misophonia Group | Emotional Dysregulation Clinical Group
Number analyzed (Participants) | 29 | 30
clusters | 0 | 0

ADVERSE EVENTS:
Time Frame: Enrollment through study completion/termination, approximately - 1-2 months.
Description: From intake through study completion, AE/SAEs, distress and risk were assessed as described in the approved DUHS IRB protocol. At the TMS visit, trained study staff queried participants on potential adverse effects that can occur during TMS pre and post TMS- including headache, neck pain, scalp pain, hearing impairment. Most of the AE reported are in relation to neurostimulation visit and only 2 other AEs, not connected to the neurostimulation visit were reported in the study.
Arm/Group | Misophonia Group | Emotional Dysregulation Clinical Group
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27
Other Adverse Events (participants affected / at risk) | 8/27 | 4/27
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Misophonia Group (N=27) | Emotional Dysregulation Clinical Group (N=27)
Headache (Nervous system disorders) | 4 (4) | 0 (0) — mild
Scalp Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) — mild
Pain (Nervous system disorders) | 1 (1) | 0 (0) — localized pain at site of TMS
Skin discomfort (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — at site of TMS neurostimulation
Eye Pain (Nervous system disorders) | 1 (1) | 0 (0) — Pain in eye that was mild which may be due to TMS frontal target engaged a nerve connected to eye.
COVID (Infections and infestations) | 0 (0) | 1 (1)
Irritability (Psychiatric disorders) | 1 (1) | 0 (0) — noise of the MRI machine made participant irritated.

LIMITATIONS AND CAVEATS:
Several protocol deviations were engaged in to accommodate participants in the study including adjusting the targeting protocol in 5 cases, imputing SUDS trial baseline values if they were left blank by participants (using the session baseline SUDS values), and adjusting intensity of stimulation for participants who found it too uncomfortable at the targeted dose.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-03-28): https://cdn.clinicaltrials.gov/large-docs/91/NCT04348591/Prot_SAP_000.pdf
  • Informed Consent Form (2022-02-04): https://cdn.clinicaltrials.gov/large-docs/91/NCT04348591/ICF_001.pdf